CLINICAL TRIAL: NCT01565512
Title: Randomized Trial to Determine the Effect of Dorsal Penile Block on Post-Robotic Prostatectomy Foley Discomfort
Brief Title: Dorsal Penile Block for Post-Robotic Prostatectomy Foley Discomfort
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding, PI left the institution, poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAI5060
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer; Robotic Prostatectomy; Foley Catheter Discomfort
Keywords: randomized trial; robotic prostatectomy; prostate cancer; foley catheter discomfort
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline injection (Placebo Comparator): saline injection
  Interventions: Drug: Saline
- Bupivacaine injection (Active Comparator): penile block with bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — A total of 100 mg bupivacaine (20 mL of 5 mg/mL solution) administered once by subcutaneous injection while patient is under general anesthesia at end of operation.
  Arms: Bupivacaine injection
Drug: Saline — A total of 20 mL on injectable saline(0.9% NS) administered once by subcutaneous injection while patient is under general anesthesia at end of operation.
  Arms: saline injection

SUMMARY:
The indwelling urethral foley is a major source of discomfort following radical prostatectomy. Our hypothesis is that intra-operative dorsal penile nerve block with bupivacaine may decrease immediate post-operative foley discomfort.

DETAILED DESCRIPTION:
Patients undergoing robot-assisted radical prostatectomy (RARP) will be randomized in a double-blind placebo controlled manner to undergo penile ring block injection at the time of skin incision closure. A visual analog scale (VAS) based questionnaire including newly developed foley discomfort scores will be administered at various time points post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* age 40 years and above,
* diagnosis of prostate cancer,
* electing to undergo robot-assisted radical prostatectomy

Exclusion Criteria:

* allergy to bupivacaine or amide-type local anesthetics,
* chronic pain condition,
* recently or currently on narcotics,
* genital abnormalities

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of pain/discomfort | postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ketan K. Badani, M.D., Principal Investigator — Assistant Professor, Department of Urology, New York Presbyterian Hospital, Columbia University Medical Center; Chris O. Wambi, M.D., Study Chair — Department of Urology, New York Presbyterian Hospital, Columbia University Medical Center; Mitchell C. Benson, M.D., Study Director — Professor and Chairman, Department of Urology, New York Presbyterian Hospital, Columbia University Medical Center
Locations (1):
- New York Presbyterian Hospital/Columbia University, New York, New York, United States